CLINICAL TRIAL: NCT00007046
Title: Genetic Study of Patients and Families With Diaphyseal Medullary Stenosis With Malignant Fibrous Histiocytoma of the Bone
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Other Study IDs: 199/15489; MTS-97-304-0001-HG; MTS-GCO-97-304HG
Record Dates: First submitted 2000-12-06; First posted 2000-12-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Stenosis; Histiocytoma
Keywords: arthritis & connective tissue diseases; bone cancer; diaphyseal medullary stenosis; genetic diseases and dysmorphic syndromes; malignant fibrous histiocytoma of bone; musculoskeletal/mesodermal cancer; oncologic disorders; rare disease
MeSH Terms: conditions — Constriction, Pathologic; Histiocytoma; Arthritis; Connective Tissue Diseases; Bone Neoplasms; Genetic Diseases, Inborn; Histiocytoma, Malignant Fibrous; Rare Diseases

SUMMARY:
OBJECTIVES: I. Identify and characterize the gene causing diaphyseal medullary stenosis with malignant fibrous histiocytoma of the bone.

II. Determine the clinical manifestations of this disease in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Blood samples are obtained from affected individuals and their family members after genetic counseling. Genetic linkage analysis is performed on these blood samples. Unaffected individuals undergo x-rays and technetium bone scans to detect the presence of bone disease. Affected individuals undergo bone densitometry, MRI studies, thallium scans, ophthalmologic examination, electrocardiogram, echocardiogram, and skin biopsies.

Affected family members identified after radiologic studies receive additional genetic counseling.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of diaphyseal medullary stenosis with malignant fibrous histiocytoma of the bone

OR

Family member, including spouses, of an affected individual

--Patient Characteristics--

Renal: Not specified

* Not pregnant
* Negative pregnancy test
* No diminished mental capacity
* No prisoners

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: J.A. Martignetti, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States